CLINICAL TRIAL: NCT04248946
Title: Sham-controlled, Double-blind, Randomised Crossover Study of the Neural, Behavioural, and Clinical Effects of Transcranial Direct Current Stimulation in Patients With a Prolonged Disorder of Consciousness; Feasibility Study
Brief Title: Neural, Behavioural, and Clinical Effects of tDCS in PDOC; Feasibility Study
Acronym: RAINDROP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Birmingham (Other)
Collaborators: Wellington Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RG_18-269
Record Dates: First submitted 2020-01-22; First posted 2020-01-30 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Consciousness Disorder; Brain Injuries; Vegetative State; Minimally Conscious State
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries; Persistent Vegetative State | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: This is a double-blind randomised crossover feasibility study of tDCS in a small cohort of PDOC individuals. The study is divided into two streams to accommodate differences in the resources available across recruitment sites: 1. MRI stream, which will include MRI and electrophysiology assessments; this is available to patients receiving care at the Wellington Hospital in London only. 2. Bedside stream, which will include electrophysiology assessments only, available to patients in specialist units at NHS (National Health Service) and non-NHS sites
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In the MRI stream all participants will receive anodal, cathodal, and sham (placebo) tDCS sessions in a randomised order. In the Bedside stream participants will receive active tDCS (either anodal or cathodal) and sham sessions also in a randomised order. A researcher not involved in data collection or analyses will programme the stimulator to deliver the specific polarity needed in each session in a double-blind manner. Sham tDCS will be delivered according to published guidelines: this mimics the physical sensations of active stimulation but does not have a neuromodulatory effect
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRI stream (Experimental): In this stream all patients receive 2 experimental interventions (anodal tDCS and cathodal tDCS) and a sham intervention (sham tDCS). These are delivered in randomised order, ensuring a balanced distribution of participants across possible orders. They will receive 5 sessions per condition (on consecutive days), for a total of 15 sessions.
  I. Anodal, cathodal, sham II. Anodal, sham, cathodal III. Cathodal, anodal, sham IV. Cathodal, sham, anodal V. Sham, anodal, cathodal VI. Sham, cathodal, anodal
  Interventions: Other: Transcranial direct current stimulation
- Bedside stream (Experimental): In this stream all patients receive 1 experimental interventions (either anodal tDCS or cathodal tDCS) and 1 sham intervention (sham tDCS). These include only 1 session per condition and are delivered in randomised order, resulting in the following possible combinations:
  I. Anodal, sham II. Cathodal, sham III. Sham, anodal IV. Sham, cathodal
  Participants will be randomly assigned to the above groups ensuring a balanced distribution of participants across them.
  Interventions: Other: Transcranial direct current stimulation

INTERVENTIONS:
Other: Transcranial direct current stimulation — tDCS alters neural excitability in a polarity-specific manner via a weak direct electric current delivered through electrodes placed on the scalp. There are 3 types of stimulation: anodal, cathodal, and sham. In anodal tDCS, the positive electrode is placed over the target brain area to increase neuronal excitability. In cathodal tDCS, the negative electrode is placed over the target brain area to decrease neuronal excitability. Sham tDCS emulates the physical sensations of active (anodal/cathodal) tDCS but current is only delivered for a short period of time and is not enough to cause any neuromodulations
  Other Names: tDCS

SUMMARY:
This study evaluates the feasibility of an experimental protocol that combines advanced multi-modal imaging of the brain with clinical and behavioural scales to characterise the neural, behavioural, and clinical effects of transcranial direct current stimulation (tDCS) for rehabilitation in PDOC

DETAILED DESCRIPTION:
Patients with prolonged disorders of consciousness (PDOC) have very limited therapeutic options, and they often show little to no progress over time. Here, the investigators will assess whether transcranial direct current stimulation can improve patients' responsiveness. The investigators will use a protocol designed to target specific brain networks that have been shown to play a key role in explaining the lack of voluntary responses in PDOC. The study will focus on characterising the mechanisms of action of tDCS and the bases for potential individual differences in responsiveness to the stimulation across participants. This feasibility study is the first step towards developing personalised tDCS interventions to restore external responsiveness in PDOC patients. Its results will inform the design of a future trial fully powered for characterising neural, behavioural, and clinical effects of tDCS in PDOC as well as the mechanisms underlying individual differences in responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Receiving care at a recruitment site, with a consensus clinical diagnosis of PDOC from any aetiology (i.e. traumatic or non-traumatic injury).
* Stable and with no need of mechanical support (i.e. respirator, etc.)

Exclusion Criteria:

* Scalp skin sores or any skin damage at the electrode sites
* Metallic implants in the face or skull
* Craniectomy or cranioplasty
* No evidence of auditory startle in clinical observations, or absent brainstem auditory evoked potentials in recent clinical history (if data available)
* MRI incompatible: metal plates incompatible with MRI scanners, pacemaker, inability to lay flat for prolonged periods of time, aneurysm clips, neurostimulators, brain/subdural electrodes, etc. (MRI stream ONLY)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Retention at end of active phase | through completion of active phase of study (tDCS intervention), on average 4 weeks for bedside stream and 8 weeks for MRI stream
  percentage of participants on study at pre-specified time points counted from the start of participation in the study (i.e., first study procedure)
Retention at 3 months | 3 months after start of participation
  percentage of participants on study at pre-specified time points counted from the start of participation in the study (i.e., first study procedure). This Outcome applies to the bedside stream only
Retention at 6 months | 6 months after start of participation
  percentage of participants on study at pre-specified time points counted from the start of participation in the study (i.e., first study procedure). This Outcome applies to the bedside stream only
Completion | through completion of active phase of study (tDCS intervention), on average 4 weeks for bedside stream and 8 weeks for MRI stream
  percentage of tDCS, MRI, and electrophysiology assessments completed per polarity

SECONDARY OUTCOMES:
Structural MRI | day 1 and day 5 of tDCS each polarity
  This will include assessments of the gross macrostructure, and microstructure of brain tissue grey matter, white matter, and cerebrospinal fluid
Functional MRI in response to task instructions | day 1 and day 5 of tDCS each polarity
  This will include assessments of the BOLD (blood oxygen level-dependent) response to characterise brain activity and connectivity during command following
EEG power in the alpha band in response to task instructions | days 1 and 4 of each polarity in the MRI stream and day 1 of each polarity in the bedside stream
  Envelope of bandpass filtered EEG data between 8-12 Hertz
EEG power in the beta band in response to task instructions | days 1 and 4 of each polarity in the MRI stream and day 1 of each polarity in the bedside stream
  Envelope of bandpass filtered EEG data between 13-30 Hertz
EMG (electromyography) amplitude changes | days 1-4 and day 2 of each polarity in the MRI and bedside streams respectively
  Changes in the amplitude of the rectified EMG signal (high-pass filtered > 50Hz) in response to instructions to move
Coma recovery scale -revised | regularly through active phase of study (baseline and outcome assessments), on average 4 weeks for bedside stream and 8 weeks for MRI stream
  clinical diagnostic scale for disorders of consciousness. Total score ranges from 0 to 23, where higher scores mean a higher level of functioning and awareness
Glasgow Outcome Scale-extended | at 3 and 6 months after start of participation
  Scale for functional outcome after brain injury. Total score ranges from 1 to 8, where higher values correspond to better outcome

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Moseley Hall Hospital, Birmingham, West Midlands
  - The Wellington Hospital, London

IPD SHARING:
Plan to Share IPD: No